CLINICAL TRIAL: NCT04617561
Title: Ursodeoxycholic Acid Combined With Low Dose Glucocorticoid in the Treatment of PBC With AIH Features II：A Randomized Controlled Open-label Clinical Trial
Brief Title: Ursodeoxycholic Acid Combined With Low Dose Glucocorticoid in the Treatment of PBC With AIH Features II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC With AIH Features II
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis, Autoimmune; Primary Biliary Cholangitis
Keywords: Glucocorticoid; Ursodeoxycholic Acid
MeSH Terms: conditions — Hepatitis, Autoimmune; Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ursodeoxycholic Acid group (Active Comparator): Ursodeoxycholic Acid 13-15mg/kg/d
  Interventions: Drug: Ursodeoxycholic acid
- Ursodeoxycholic Acid+Low Dose Glucocorticoid group (Experimental): Ursodeoxycholic Acid 13-15mg/kg/d+Methylprednisolone 12mg/d in induction period and 2-4mg/d in maintenance period
  Interventions: Drug: Ursodeoxycholic acid+Low Dose Glucocorticoid(Methylprednisolone)

INTERVENTIONS:
Drug: Ursodeoxycholic acid — Participants received Ursodeoxycholic acid (13-15mg/kg/d po.)
  Other Names: UDCA;Ursofalk(250mg*25,Losan Pharma GmbH)
  Arms: Ursodeoxycholic Acid group
Drug: Ursodeoxycholic acid+Low Dose Glucocorticoid(Methylprednisolone) — Participants received Methylprednisolone (12mg/d po. in induction and 2-4mg/d in maintenance) combined with Ursodeoxycholic acid (13-15mg/kg/d po.)
  Other Names: Medrol（4mg*30,pfizer ltalia srl)
  Arms: Ursodeoxycholic Acid+Low Dose Glucocorticoid group

SUMMARY:
A randomized controlled open-label clinical trial of ursodeoxycholic acid combined with low dose glucocorticoid in the treatment of PBC With AIH Features II to asses efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years;
2. The diagnosis of PBC is clear and does not meet the Paris criteria for diagnosing PBC overlap AIH, but it needs to meet 3xULN < ALT < 5xULN or 3xULN < AST < 5xULN or 1.3xULN < IgG < 2xULN, and liver pathological biopsy excludes moderate or higher interface inflammation;
3. Agreed to participate in the trial, and assigned informed consent.

Exclusion Criteria:

1. The presence of hepatitis A, B, C, D, or E virus infection;
2. Patients with presence of cirrhosis;
3. Patients with presence of fulminant liver failure;
4. Liver damage caused by other reasons: such as primary sclerosing cholangitis, non-alcoholic steatohepatitis, drug induced liver disease or Wilson's disease; Pregnant and breeding women and women of childbearing age in need of reproduction;
5. Severe disorders of other vital organs, such as severe heart failure, cancer;
6. Parenteral administration of blood or blood products within 6 months before screening;
7. Recent treatment with drugs having known liver toxicity;
8. Taken part in other clinic trials within 6 months before enrollment.
9. patients with contraindications of glucocorticoid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission | up to 12 months
  The percentage of patients in biochemical remission, defined as normalization of serum ALT and IgG levels after treatment, per treatment group.

SECONDARY OUTCOMES:
Partial remission | up to 12 months
  Partial remission, defined as ALT or AST serum levels >1x Upper Limit of Normal (ULN) and <2x ULN
Minimal response | up to 12 months
  Minimal response, defined as decrease of ALT or AST serum levels but still >2x ULN
Treatment failure | up to 12 months
  defined as no improvement or increase of ALT or AST serum levels
ALT,AST,IgG | baseline and month 3,6,12
  serum ALT,AST and IgG levels
percentage of immune cells | baseline and month 12
  percentage of T cells, cDC, MDSC, Treg, Breg, plasma cells, NK, NKT
Side-effects | up to 12 months
  Drug related side-effects

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology & Hepatology,West China Hospital,Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No